CLINICAL TRIAL: NCT00001723
Title: Safety and Efficacy of Orlistat (Xenical, Hoffmann LaRoche) in African American and Caucasian Children and Adolescents With Obesity-Related Comorbid Conditions
Brief Title: Safety and Efficacy of Xenical in Children and Adolescents With Obesity-Related Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jack Yanovski (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Jack Yanovski, Section Chief, Section on Growth and Obesity, PDEGEN, NICHD, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 980111; 98-CH-0111 (Other: NICHD IRB)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2012-12-18 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Mellitus; Hypertension; Metabolic Disease; Obesity; Sleep Apnea Syndrome
Keywords: Dyslipidemia; Race; Body Fat; Visceral Fat; Sleep Apnea; Fat-Soluble Vitamins; Type 2 Diabetes; Obesity; Childhood Obesity
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Metabolic Diseases; Obesity; Sleep Apnea Syndromes; Dyslipidemias; Diabetes Mellitus, Type 2; Pediatric Obesity | interventions — Orlistat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo 120 mg TID x 6 months plus a behavioral weight loss program
  Interventions: Drug: Placebo
- Orlistat (Experimental): Orlistat 120 mg TID for 6 months plus a behavioral weight loss program
  Interventions: Drug: Orlistat

INTERVENTIONS:
Drug: Orlistat — Subjects receive drug for 6 months plus a 12 week intensive behavioral weight los program. Subjects return for monthly visits for 3 more months.
  Other Names: Xenical (orlistat)capsules
  Arms: Orlistat
Drug: Placebo — Subjects receive drug for 6 months plus a 12 week intensive behavioral weight los program. Subjects return for monthly visits for 3 more months.
  Other Names: Placebo capsule
  Arms: Placebo

SUMMARY:
Obesity is a condition affecting one-third off the U.S. population and is a major risk actor for the development of Type 2 diabetes, hyperlipidemia (increased levels of fat in the blood), hypertension (high blood pressure), and other disorders of the heart and lungs. Individuals with the onset of obesity during childhood or adolescence are at an increased risk of obesity-related, diseases, both during adolescence and later in adult life.

African American girls and women are at an increased risk for obesity, and have substantial rates of obesity-related diseases and causes of death. Further, many African American adult women fail to respond to many of the therapeutic approaches used to treat obesity. At present there are no medical therapies proven effective for the correction of severe obesity in children or adolescents.

One medication that may have a favorable risk-benefit ratio in pediatric populations is Orlistat (Xenical, Hoffmann LaRoche). Orlistat works by preventing the action of enzymes in the digestive process, interfering with the absorption of approximately 1/3 of the fat eaten in the diet. Xenical appears to be effective for reducing weight and obesity-associated diseases in obese adults.

Researchers propose to determine the safety, tolerability, and efficacy of Xenical in 12-17 year old severely obese African American and Caucasian children and adolescents who have one or more obesity-related disease (hypertension, hyperlipidemia, sleep apnea, hepatic steatosis, insulin resistance, impaired glucose tolerance, or Type 2 diabetes).

DETAILED DESCRIPTION:
Obesity is a condition affecting one-third of the adult U.S. population and is a major risk factor for the development of Type 2 diabetes, hyperlipidemia, hypertension, and other cardiovascular and respiratory disorders. Individuals with the onset of obesity during childhood or adolescence are at increased risk for obesity-related, comorbid conditions, both during adolescence and later in life. African American girls and women are at particular risk for obesity, and have substantial rates of obesity-related morbidity and mortality. Further, African American adult women have a less satisfactory response to many therapeutic approaches used to treat obesity. At present, there are no medical therapies proven effective for the amelioration of severe obesity in children or adolescents. One medication that may have a favorable risk-benefit ratio in pediatric populations is orlistat (Xenical(Trademark), Hoffmann LaRoche). Orlistat acts by inhibiting gastrointestinal lipases, interfering with the absorption of approximately 1/3 of ingested dietary fat. Orlistat appears to be effective for reducing weight and obesity-associated comorbidities in obese adults. We propose to determine the safety, tolerability, and efficacy of orlistat in 12-17 year-old severely obese African American and Caucasian children and adolescents who have one or more obesity-related comorbidity (hypertension, hyperlipidemia, sleep apnea, hepatic steatosis, insulin-resistance, impaired glucose tolerance, or Type 2 diabetes). Under this protocol, we have conducted an open-label pilot study of orlistat in twenty subjects, suggesting orlistat has a similar side effect profile in adolescents as in adults. We wish to determine the safety and efficacy of orlistat in reducing obesity-related comorbidities using a randomized, double-blind, placebo-controlled clinical trial. All study participants will be enrolled in a psycho-educational weight loss program that includes nutrition education, cognitive-behavioral self-monitoring strategies, and promotion of physical activity. We will also study the effects of orlistat on fat preferences, and study the influence of genetic variables on energy expenditure and weight loss during treatment. A group of healthy, non-overweight children and adolescents will complete questionnaires and exercise studies as a control group for interpretation of results in overweight children and adolescents, but will not undergo phlebotomy or receive any medication.

ELIGIBILITY:
* INCLUSION CRITERIA:

Good general health. Individuals taking medications for obesity-related comorbid conditions will not be excluded.

Obesity: body mass index for age and triceps skinfold above the 95th percentile (determined by NHANES I age-, sex-, and race- specific data). All subjects will be required to be over 60 kg in body weight.

Evidence for a quantifiable obesity-related comorbidity. Examples include: systolic or diastolic hypertension (determined by age-specific charts); frank Type 2 diabetes, impaired glucose tolerance assessed by oral glucose tolerance testing; hyperinsulinemia (defined as a fasting insulin greater than 15 mIU/mL); significant hyperlipidemia (total cholesterol greater than 200 mg/dL, LDL cholesterol greater than 129 mg/dL or fasting triglycerides greater than 200 mg/dL); hepatic steatosis (SGPT or SGOT above normal range with negative hepatitis studies) or sleep apnea documented by a sleep study.

Age 12 to 17 years at the start of the study.

For girls with childbearing potential, a negative pregnancy test before taking and while taking study medication. Sexually active females must be using an effective form of birth control. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonogestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these cannot be used, contraceptive foam with a condom is recommended.

Race of all four grandparents self-identified as either all Caucasian or all African American.

EXCLUSION CRITERIA:

Volunteers will be excluded (and referred to non-experimental treatment programs) for the following reasons:

Presence of renal, hepatic (other than obesity-related steatosis), gastrointestinal, most endocrinologic (e.g., Cushing syndrome), or pulmonary disorders (other than either asthma not requiring continuous medication or sleep apnea-related disorders);

Adolescent girls who are pregnant, who are currently nursing an infant, or who are having unprotected intercourse;

Individuals who have, or whose parent or guardians have, current substance abuse or a psychiatric disorder or other condition which, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study;

Subjects who regularly use prescription medications unrelated to the complications of obesity. Oral contraceptive use will be permitted, provided the contraceptive has been used for at least two months before starting study medication. The use of over-the-counter and prescription medications will be reviewed on a case-by-case basis; depending on the medication, subjects who have continued to take prescription medication for at least 3 months prior to study entry may be eligible;

Recent use (within six months) of anorexiant medications for the purpose of weight reduction;

Inability to undergo MRI (e.g., volunteers with metal within their bodies including cardiac pacemakers, neural pacemakers, aneurysmal clips, shrapnel, ocular foreign bodies, cochlear implants, non-detachable electronic or electromechanical devices such as infusion pumps, nerve stimulators, bone growth stimulators, etc. that are contraindications).

For pilot study participants, hypersensitivity or allergy to methylene blue. Individuals with documented G6PD deficiency will be excluded.

INCLUSION CRITERIA: HEALTHY CONTROL CHILDREN AND ADOLESCENTS:

Volunteers will qualify for inclusion if they meet the following criteria:

1. Good general health.
2. Age 12-17 years at study entry.
3. Body mass index (BMI) for age above the 5th percentile and below 85th percentile, which is considered normal weight by CDC growth chart standards.
4. For females with childbearing potential, a negative pregnancy test at initial evaluation.
5. Race of all four grandparents self-identified as either all Caucasian or all African American.

EXCLUSION CRITERIA: HEALTHY CONTROL CHILDREN AND ADOLESCENTS:

Volunteers will be excluded for the following reasons:

1. Presence of past or present medical problems which would impair performance during the exercise tests;
2. Females who are pregnant, or who are currently nursing an infant;
3. Individuals who have, or whose parent or guardian has, current substance abuse or a psychiatric disorder or other condition that in the opinion of the investigators would impede competence or possibly hinder completion of the study;
4. Recent weight change of more than 3% of body weight in the past two months;
5. Recent use (within six months) of anorexiant medications for the purpose of weight reduction;
6. Physical impairments that would prevent completion of either the walk/run test or the cycle test.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 1998-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kuczmarski RJ, Flegal KM, Campbell SM, Johnson CL. Increasing prevalence of overweight among US adults. The National Health and Nutrition Examination Surveys, 1960 to 1991. JAMA. 1994 Jul 20;272(3):205-11. doi: 10.1001/jama.272.3.205. PMID 8022039
- [Background] Drent ML, Larsson I, William-Olsson T, Quaade F, Czubayko F, von Bergmann K, Strobel W, Sjostrom L, van der Veen EA. Orlistat (Ro 18-0647), a lipase inhibitor, in the treatment of human obesity: a multiple dose study. Int J Obes Relat Metab Disord. 1995 Apr;19(4):221-6. PMID 7627244
- [Background] Must A, Jacques PF, Dallal GE, Bajema CJ, Dietz WH. Long-term morbidity and mortality of overweight adolescents. A follow-up of the Harvard Growth Study of 1922 to 1935. N Engl J Med. 1992 Nov 5;327(19):1350-5. doi: 10.1056/NEJM199211053271904. PMID 1406836
- [Background] Chanoine JP, Hampl S, Jensen C, Boldrin M, Hauptman J. Effect of orlistat on weight and body composition in obese adolescents: a randomized controlled trial. JAMA. 2005 Jun 15;293(23):2873-83. doi: 10.1001/jama.293.23.2873. PMID 15956632
- [Result] McDuffie JR, Calis KA, Uwaifo GI, Sebring NG, Fallon EM, Frazer TE, Van Hubbard S, Yanovski JA. Efficacy of orlistat as an adjunct to behavioral treatment in overweight African American and Caucasian adolescents with obesity-related co-morbid conditions. J Pediatr Endocrinol Metab. 2004 Mar;17(3):307-19. doi: 10.1515/jpem.2004.17.3.307. PMID 15112907
- [Result] McDuffie JR, Calis KA, Booth SL, Uwaifo GI, Yanovski JA. Effects of orlistat on fat-soluble vitamins in obese adolescents. Pharmacotherapy. 2002 Jul;22(7):814-22. doi: 10.1592/phco.22.11.814.33627. PMID 12126214
- [Result] McDuffie JR, Calis KA, Uwaifo GI, Sebring NG, Fallon EM, Hubbard VS, Yanovski JA. Three-month tolerability of orlistat in adolescents with obesity-related comorbid conditions. Obes Res. 2002 Jul;10(7):642-50. doi: 10.1038/oby.2002.87. PMID 12105286
- [Derived] Omotosho YB, Reynolds JC, Yanovski JA, Tatsi C. Body Composition and Fat Deposition in Children with Cushing Disease and Associations with Cardiometabolic Risk Factors. J Pediatr. 2025 Dec 3;290:114933. doi: 10.1016/j.jpeds.2025.114933. Online ahead of print. PMID 41349930
- [Derived] Schvey NA, Shank LM, Tanofsky-Kraff M, Ramirez S, Altman DR, Swanson T, Rubin AG, Kelly NR, LeMay-Russell S, Byrne ME, Parker MN, Broadney MM, Brady SM, Yanovski SZ, Yanovski JA. Weight-based teasing in youth: Associations with metabolic and inflammatory markers. Pediatr Obes. 2021 Mar;16(3):e12729. doi: 10.1111/ijpo.12729. Epub 2020 Oct 15. PMID 33059389
- [Derived] Han JC, Reyes-Capo DP, Liu CY, Reynolds JC, Turkbey E, Turkbey IB, Bryant J, Marshall JD, Naggert JK, Gahl WA, Yanovski JA, Gunay-Aygun M. Comprehensive Endocrine-Metabolic Evaluation of Patients With Alstrom Syndrome Compared With BMI-Matched Controls. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2707-2719. doi: 10.1210/jc.2018-00496. PMID 29718281
- [Derived] Radin RM, Tanofsky-Kraff M, Shomaker LB, Kelly NR, Pickworth CK, Shank LM, Altschul AM, Brady SM, Demidowich AP, Yanovski SZ, Hubbard VS, Yanovski JA. Metabolic characteristics of youth with loss of control eating. Eat Behav. 2015 Dec;19:86-9. doi: 10.1016/j.eatbeh.2015.07.002. Epub 2015 Jul 18. PMID 26210388
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1998-CH-0111.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual for RCT began in 1999 and ended in 2008. All subjects were screened at the NIH Clinical Center.
Pre-assignment Details: Most subjects screened but not enrolled (101) did not have an obesity-related comorbid condition (i.e., hypertension or dyslipidemia). 16 met a medical exclusion, and 13 declined participation after undergoing initial evaluation.
Groups:
- Orlistat: Orlistat 120 mg TID for 6 months plus a behavioral weight loss program
  Orlistat : Subjects receive drug for 6 months plus a 12 week intensive behavioral weight los program. Subjects return for monthly visits for 3 more months.
- Placebo: Matching placebo 120 mg TID x 6 months plus a behavioral weight loss program
  Placebo : Subjects receive drug for 6 months plus a 12 week intensive behavioral weight los program. Subjects return for monthly visits for 3 more months.
Period: Overall Study
Arm/Group | Orlistat | Placebo
Started | 100 | 100
Completed | 87 | 84
Not Completed | 13 | 16
Not completed — Lack of Efficacy | 6 | 7
Not completed — Lack of family interest | 4 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — medication intolerance | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Orlistat | Placebo | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100 | 100 | 200
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 14.65 (1.38) | 14.52 (1.46) | 14.59 (1.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 66 | 131
  Male | 35 | 34 | 69
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Change in BMI Standard Deviation Score
Description: Body Mass index standard deviation score calculated for age and sex according to Centers for Disease Control standards. See: Kuczmarski RJ, Ogden CL, Guo SS, Grummer-Strawn LM, Flegal KM, Mei Z et al. 2000 CDC Growth Charts for the United States: methods and development. Vital Health Stat 11 2002; (246): 1-190.
Time Frame: baseline to 6 months
Population: Multiple imputation analysis
Measure: Mean (Standard Error); unit: Standard Deviation Score
Arm/Group | Orlistat | Placebo
Number analyzed (Participants) | 100 | 100
Standard Deviation Score | -0.12 (0.02) | -0.06 (0.02)
Statistical Analysis 1: Comparison: Orlistat vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA

2. Secondary Outcome: Change in Body Weight
Description: Weight in kg
Time Frame: baseline to 6 months
Population: Multiple imputation analysis
Measure: Mean (Standard Error); unit: kg
Arm/Group | Orlistat | Placebo
Number analyzed (Participants) | 100 | 100
kg | -2.9 (0.7) | -0.6 (0.7)

3. Secondary Outcome: Change in Body Mass Index
Description: BMI is calculated in kg/m2. Change from baseline to 6 months of treatment
Time Frame: baseline to 6 months
Population: Muliple imputation analysis
Measure: Mean (Standard Error); unit: kg per square meter
Arm/Group | Orlistat | Placebo
Number analyzed (Participants) | 100 | 100
kg per square meter | -1.44 (0.26) | -0.50 (0.20)

4. Secondary Outcome: Change in Body Fat (kg)
Description: body fat distribution measures obtained from Dual-energy X-ray Absorptiometry (DEXA)
Time Frame: baseline to 6 months
Population: Multiple Imputation analysis
Measure: Mean (Standard Error); unit: kg
Arm/Group | Orlistat | Placebo
Number analyzed (Participants) | 100 | 100
kg | -3.2 (0.55) | -1.7 (0.53)

5. Secondary Outcome: Effect of Race on Change in Weight (kg)
Description: Difference in change of weight in kg according to race (Non-Hispanic White versus Non-Hispanic Black)
Time Frame: baseline to 6 months
Population: Multiple imputation analysis
Measure: Mean (Standard Error); unit: kg
Groups:
- Orlistat - Non-Hispanic Blacks: Change in weight for Non-Hispanic Black participants treated with orlistat
- Orlistat - Non- Hispanic Whites: Change in weight for Non-Hispanic White participants treated with orlistat
- Placebo - Non-Hispanic Blacks: Change in weight for Non-Hispanic Black participants treated with placebo
- Placebo - Non-Hispanic Whites: Change in weight for Non-Hispanic White participants treated with placebo
Arm/Group | Orlistat - Non-Hispanic Blacks | Orlistat - Non- Hispanic Whites | Placebo - Non-Hispanic Blacks | Placebo - Non-Hispanic Whites
Number analyzed (Participants) | 63 | 37 | 60 | 40
kg | -2.126 (0.812) | -3.742 (1.046) | 0.415 (0.835) | -1.580 (1.013)

ADVERSE EVENTS:
Time Frame: 6 months of randomized treatment
Arm/Group | Orlistat | Placebo
Serious Adverse Events (participants affected / at risk) | 0/100 | 2/100
Other Adverse Events (participants affected / at risk) | 95/100 | 94/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Orlistat (N=100) | Placebo (N=100)
Hypoglycemia - pharmacy error in preparing insulin (Endocrine disorders) | 0 | 1
Left lower quadrant pain and vomiting - admitted overnight (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Orlistat (N=100) | Placebo (N=100)
ear disorders (otitis, earache, ear pain) (Ear and labyrinth disorders) | 7 | 7
eye disorders (change in vision, conjunctivitis, styes) (Eye disorders) | 8 | 9
abdominal pain or cramping (Gastrointestinal disorders) | 16 | 21
bloating or gas (Gastrointestinal disorders) | 18 | 5
BORBORYGMI (Gastrointestinal disorders) | 6 | 2
constipation (Gastrointestinal disorders) | 1 | 7
Controlled discharge of oil without stool (Gastrointestinal disorders) | 56 | 11
Decreased frequency of bowel movements (Gastrointestinal disorders) | 25 | 22
diarrhea (Gastrointestinal disorders) | 21 | 8
fatty-appearing stools (Gastrointestinal disorders) | 61 | 6
flatulence (passage of gas) (Gastrointestinal disorders) | 60 | 47
flatus with discharge (Gastrointestinal disorders) | 43 | 11
frequent urge for bowel movement (Gastrointestinal disorders) | 19 | 3
hiccups (Gastrointestinal disorders) | 1 | 3
Increased frequency of bowel movements (Gastrointestinal disorders) | 68 | 45
NAUSEA (Gastrointestinal disorders) | 10 | 9
oily spotting (Gastrointestinal disorders) | 6 | 0
rectal bleeding - hemorrhoids (Gastrointestinal disorders) | 4 | 2
soft or deliquescent stools (Gastrointestinal disorders) | 68 | 42
stomach pain or cramps (Gastrointestinal disorders) | 8 | 9
Stools almost all liquid with very few solid parts (Gastrointestinal disorders) | 64 | 34
Stools hard and in the shape of small pellets (Gastrointestinal disorders) | 11 | 10
Stools mixed with fat or with a separate oily layer (Gastrointestinal disorders) | 83 | 18
uncontrolled passage of stool or oil (Gastrointestinal disorders) | 60 | 11
Urgent, but controlled, need to produce stools (Gastrointestinal disorders) | 44 | 18
Vomiting (Gastrointestinal disorders) | 7 | 7
dizziness (General disorders) | 4 | 4
epistaxis (General disorders) | 5 | 2
feeling cold (General disorders) | 5 | 2
headache (General disorders) | 14 | 17
increased sweating (General disorders) | 3 | 4
increased thirst (General disorders) | 5 | 4
sinusitis, post-nasal drip or nasal stuffiness (General disorders) | 2 | 5
unusual tiredness or weakness (fatigue) (General disorders) | 1 | 5
Pharyngitis (Infections and infestations) | 6 | 12
sinusitis, post-nasal drip or nasal stuffiness (Infections and infestations) | 1 | 3
decrease in appetite (Metabolism and nutrition disorders) | 11 | 9
muscle pain, stiffness, cramps, or ache (Musculoskeletal and connective tissue disorders) | 16 | 12
migraine headaches (Nervous system disorders) | 3 | 0
mental depression (Psychiatric disorders) | 1 | 3
dysuria or UTI (Renal and urinary disorders) | 1 | 5
nocturia (Renal and urinary disorders) | 0 | 3
Asthma symptoms (Respiratory, thoracic and mediastinal disorders) | 5 | 3
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 14 | 17
skin rash (Skin and subcutaneous tissue disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes